CLINICAL TRIAL: NCT05663411
Title: An Open-label, Randomized, Active-Controlled Dose Titration Study to Assess the Efficacy and Safety of SHR6508 in Hemodialysis Subjects With Secondary Hyperparathyroidism
Brief Title: A Study of SHR6508 in Secondary Hyperparathyroidism
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR6508-201
Record Dates: First submitted 2022-12-14; First posted 2022-12-23 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2022-11

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — Cinacalcet

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A: SHR6508 (Experimental)
  Interventions: Drug: SHR6508
- Treatment group B: SHR6508 (Experimental)
  Interventions: Drug: SHR6508
- Treatment group C: Cinacalcet (Active Comparator)
  Interventions: Drug: Cinacalcet

INTERVENTIONS:
Drug: SHR6508 — SHR6508
  Arms: Treatment group A: SHR6508
Drug: SHR6508 — SHR6508
  Arms: Treatment group B: SHR6508
Drug: Cinacalcet — Cinacalcet
  Arms: Treatment group C: Cinacalcet

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR6508 for Chinese patients with secondary hyperparathyroidism of chronic kidney disease treated by maintenance hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Diagnosed with end stage renal disease receiving stable hemodialysis
3. Male or female
4. Meet the Body Mass Index standard
5. Stably use of concomitant medication of other therapies of SHPT
6. Meet the standard of iPTH level, cCa and HB

Exclusion Criteria:

1. Subjects with a history of malignant tumor
2. Subjects with neuropsychiatric diseases
3. Subjects with a history of cardiovascular diseases
4. Subjects with gastrointestinal diseases
5. Subjects with a history of surgery
6. Subjects with a history of blood loss
7. Subjects with a history of kidney transplant
8. Abnormal blood pressure, serum magnesium, serum transaminase, serum albumin
9. Subjects with a treatment history of similar drugs
10. Allergic to a drug ingredient or component
11. Pregnant or nursing women
12. No birth control during the specified period of time
13. Subject with a history of alcohol abuse and drug abuse
14. Participated in clinical trials of other drugs
15. The investigators determined that other conditions were inappropriate for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in serum iPTH | Baseline and the efficacy period, defined as Week 16
  iPTH was tested at a central laboratory.

SECONDARY OUTCOMES:
Proportion of Participants to End of Study whose iPTH decreased by≥30% from baseline | Baseline and the efficacy period, defined as Week 16
  iPTH was tested at a central laboratory.
Proportion of Participants to End of Study whose iPTH decreased to 300 pg/mL from baseline | Baseline and the efficacy period, defined as Week 16
  iPTH was tested at a central laboratory.
Change From Baseline in serum cCa and P | Baseline and the efficacy period, defined as Week 16
  cCa and P were tested at a local laboratory.
Participants With Treatment-Emergent Adverse Events (TEAEs) | Day1 to End of Study, End of Study is about Week 20
  Terms were coded with Medical Dictionary for Regulatory Activities (MedDRA)
Participants with Anti-SHR6508 Antibody at baseline and postbaseline | Day1 to End of Study, End of Study is about Week 20

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided